CLINICAL TRIAL: NCT07255677
Title: Effect of Stretching Exercises Versus Aerobic Exercises on Preeclampsia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Khaled Abdrabo Naeem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005974
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching exercises program + Antihypertensive drugs (Experimental): It will consist of 30 women with mild preeclampsia. They will be treated with a stretching exercise program, conducted three times per week for six weeks, alongside antihypertensive drugs.
  Interventions: Other: Stretching exercises program; Drug: Antihypertensive drugs
- Aerobic exercises program + Antihypertensive drugs (Experimental): It will consist of 30 women with mild preeclampsia. They will be treated with an aerobic exercise program, conducted three times per week for six weeks, alongside antihypertensive drugs.
  Interventions: Other: Aerobic exercises program; Drug: Antihypertensive drugs

INTERVENTIONS:
Other: Stretching exercises program — Each woman in the first experimental group will follow a supervised stretching exercise program three times per week for six weeks. Sessions will begin with deep breathing warm-up, followed by stretching each target muscle for 10 seconds with 10 seconds relaxation for the first two weeks, 15 seconds stretching and relaxation in weeks three and four, and 20 seconds in weeks five and six. Each stretch will be repeated 10 times per session. After six weeks, women will be instructed to continue these exercises until delivery.
  Arms: Stretching exercises program + Antihypertensive drugs
Other: Aerobic exercises program — The second experimental group will follow a supervised aerobic exercise program of mild to moderate intensity (40%-60% HRmax, calculated as 220 minus age). Heart rate will be monitored before and during exercise. The program, conducted three times per week for six weeks, will start with a 5-minute low-speed walking warm-up. In the first two weeks, this will be followed by 10 minutes on a treadmill (King Fitness Model 8000AC), 5 minutes relaxation, 10 minutes on a stationary bike (GRASP93026), and 5 minutes relaxation. In weeks three and four, treadmill and bike sessions will increase to 15 minutes each, with 10 minutes relaxation between. In weeks five and six, treadmill and bike time will increase to 20 minutes, with 15 minutes relaxation between. After six weeks, women will continue these exercises until delivery.
  Arms: Aerobic exercises program + Antihypertensive drugs
Drug: Antihypertensive drugs — All women in both groups will be treated by antihypertensive drugs (labipress) for 6 weeks.
  Other Names: labipress

SUMMARY:
The purpose of the study is to compare between the effect of stretching exercises and aerobic exercises on preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia increases maternal morbidity and mortality since the 1980s, Studies from the World Health Organization also showed an increased risk of hemorrhagic stroke with history of hypertension in pregnancy. In addition to this increased risk of thrombosis, there is also increased morbidity and mortality associated specifically with stroke in these women. PE lead to preterm delivery and increase neonatal morbidity such as Intrauterine Growth Restriction (IUGR), Risk of Fet al Demise/Stillbirth, and infants have a nine times greater incidence of respiratory distress syndrome than full-term neonate.

Medical treatments of preeclampsia . have a lot of side effects on mother and fetus. So, we are going to study more effective noninvasive therapy methods to prevent and decrease the risk of PE. In this randomized controlled study (RCT).

Several studies have explored the impact of exercise on the management and prevention of preeclampsia:

The Effect of Maternal Exercise Program on Fet al Growth in Pre-Eclampsia: A Prospective, Randomized Controlled Clinical Trial investigated the impact of a structured maternal exercise program on fet al growth in women diagnosed with preeclampsia. The findings suggested that regular, supervised exercise could positively influence fet al growth parameters in this cases. Impact of Exercise Training on Preeclampsia: Potential Preventive Mechanisms This review examined the potential mechanisms through which exercise training might reduce the risk of developing preeclampsia. The authors discussed how regular physical activity could improve endothelial function, reduce oxidative stress, and modulate immune responses, thereby potentially lowering preeclampsia risk. Aerobic Exercise Training in Formerly Preeclamptic Women: Effects on Venous Reserve In this study, they examined the effects of aerobic exercise training on venous reserves in 24 normotensive formerly preeclamptic women and 20 controls. Before and after 12-week aerobic exercise training, they demonstrate that 12 weeks of aerobic exercise training effectively improves venous reserve capacity in postpartum women. An umbrella review by Martínez highlighted that prenatal exercise can lead to systolic blood pressure (SBP) reductions of about 9.6 mmHg, alongside significant reductions in diastolic blood pressure (DBP) - with substantial evidence quality. In 2023 a meta-analysis of 14 RCTs (2010-2023) confirmed that prenatal physical activity reduces the risk of gestational hypertensive disorders by 56% and lowers SBP by 2.64 mmHg and DBP by 1.99 mmHg. More specifically, a meta-analysis focusing on aerobic and resistance training showed that while exercise didn't significantly change BP in low-risk pregnancies, in at-risk women it reduced SBP by 3.91 mmHg and DBP by 2.9 mmHg.

Another meta-analysis of 18 RCTs reported overall mean reductions of SBP by 3.19 mmHg and DBP by 2.14 mmHg in exercising pregnant women compared to controls.

Comparing studies like study done by Awad 2019 to find Effect of stretching exercises versus autogenic training on preeclampsia research published in the Journal of Advanced Pharmaceutical Technology & Research compared the effects of stretching exercises and autogenic training on preeclamptic women. The study found that both interventions led to significant reductions in blood pressure and proteinuria levels, with stretching exercises showing a slightly more pronounced effect. This indicates that stretching can be an effective non-pharmacological approach to managing preeclampsia symptoms, another comparison of walking versus stretching exercises to reduce the incidence of preeclampsia: a randomized clinical trial a study conducted by the University of North Carolina at Chapel Hill found that pregnant women with a history of preeclampsia who engaged in regular stretching exercises experienced a lower incidence of the condition compared to those who participated in walking programs. Specifically, 5% of women in the stretching group developed preeclampsia, versus 14% in the walking group. The researchers hypothesized that stretching might increase levels of transferrin, a protein that combats oxidative stress, thereby offering protective benefits.

ELIGIBILITY:
Inclusion Criteria:

* Their ages ranged from 20-30 years old.
* Their body mass index (BMI) didn't exceed 35 Kg\m2.
* All women primigravida.
* All women are complaining of mild preeclampsia.

Exclusion Criteria:

* Chronic disease (diabetes mellitus, thyroid, hypertension, nephrotic).
* Vaginal bleeding.
* Placenta previa.
* Physical and psychological disorders.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of arterial blood pressure | 6 weeks
  Arterial blood pressure will be measured from the right arm while the woman is in a half-lying position. The measurement will be the mean of three trials. Each woman in both groups will be assessed before and after the six-week treatment period.
Measurement of proteinuria | 6 weeks
  Each woman in both groups will be asked to collect a 24-hour urine sample in sterilized glass bottles for measurement of protein levels. This collection will take place before and after the six-week treatment period.

SECONDARY OUTCOMES:
Body mass index (BMI) measurement | 6 weeks
  The BMI of each woman in both groups will be calculated before and after treatment with this calculation:
  Body mass index (BMI)= Weight (Kg) / Height (m2).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmad Mohamed Awad, PhD, Study Chair — Professor, Cairo university; Mai Mohamed Ali, PhD, Study Director — Assistant Professor, Cairo University; Amir Araby Gabre, PhD, Study Director — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt